CLINICAL TRIAL: NCT01984606
Title: A Phase IIIb Randomised, Double-blind, Active-controlled, Parallel Group, Efficacy and Safety Study of Once Daily Oral Administration of Empagliflozin 25 mg Compared to Sitagliptin 100 mg During 52 Weeks in Type 2 Diabetes Mellitus Patients Who Are Treatment-naïve or on Treatment With Metformin With Insufficient Glycaemic Control
Brief Title: Efficacy and Safety of Empagliflozin Versus Sitagliptin in Patients With Type 2 Diabetes
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1245.22; 2013-000060-29 (EudraCT Number: EudraCT)
Record Dates: First submitted 2013-11-08; First posted 2013-11-14 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin; Sitagliptin Phosphate

ARMS (2):
- Empagliflozin (Experimental): Empagliflozin once daily
  Interventions: Drug: Empagliflozin; Drug: Placebo
- Sitagliptin (Active Comparator): Sitagliptin once daily
  Interventions: Drug: Sitagliptin; Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin — Empagliflozin once daily
  Arms: Empagliflozin
Drug: Placebo — Placebo matching empagliflozin
  Arms: Empagliflozin
Drug: Sitagliptin — Sitagliptin once daily
  Arms: Sitagliptin
Drug: Placebo — Placebo matching sitagliptin
  Arms: Sitagliptin

SUMMARY:
The purpose of this study is to assess safety and efficacy of empagliflozin compared to sitagliptin in patients with type 2 diabetes mellitus who are treatment-naive or on treatment with metformin and have insufficient glycaemic control. The study will assess non-inferiority of empagliflozin to sitagliptin with regards to HbA1c.

ELIGIBILITY:
Inclusion criteria:

Inclusion criteria:

* Diagnosis of type 2 diabetes mellitus.
* Male and female patients on diet and exercise regimen who are:
* Treatment-naïve, defined as absence of any oral antidiabetic therapy for 12 weeks prior to randomisation.

or

* Pre-treated with immediate release metformin unchanged for 10 weeks prior to randomisation. Minimum dose for metformin: >=1500 mg/day or maximum tolerated dose or maximum dose according to local label.
* HbA1c of >= 7.5 % and <= 10.5 % at Visit 1 and 3.
* Age >= 18 yrs.

Exclusion criteria:

* Uncontrolled hyperglycaemia with a glucose level >270 mg/dL (>15 mmol/L) after an overnight fast during dose stabilisation (if applicable) and/or placebo run-in.
* Any other antidiabetic drug within 12 weeks prior to randomisation (applicable to treatment-naïve patients).
* Any other antidiabetic drug within 10 weeks prior to randomisation except metformin (applicable to patients on background treatment with metformin).
* Acute coronary syndrome (non-STEMI, STEMI and unstable angina pectoris), stroke or TIA within 3 months prior to informed consent.
* Indication of liver disease.
* Moderate to severe renal impairment.
* Bariatric surgery within the past two years.
* Treatment with anti-obesity drugs 3 months prior to informed consent.
* Current treatment with systemic steroids at time of informed consent or any other uncontrolled endocrine disorder except type 2 diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
The change from baseline in HbA1c after 52 weeks of treatment. | Baseline and week 52

SECONDARY OUTCOMES:
The change in bodyweight (kg) from baseline after 52 weeks of treatment | Baseline and week 52
The change in Systolic Blood Pressure (SBP) from baseline after 52 weeks of treatment | Baseline and week 52
The coefficient of durability of HbA1c response between 24 weeks and 52 weeks of treatment | Week 24 and week 52
The change in Diastolic Blood Pressure (DBP) from baseline after 52 weeks of treatment | Baseline and week 52

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim